CLINICAL TRIAL: NCT03605797
Title: Fixation of Sacral Fractures by Posterior Tension Band Plating
Brief Title: Fixation of Sacral Fractures by Posterior Plate
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaaeldin Mohamed Abdelhafez, Principal Investigator, Assiut University
Other Study IDs: TBP
Record Dates: First submitted 2018-07-11; First posted 2018-07-30 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Sacral Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No intervention: To study the indication and results of fixing the sacral fracture by tension band plating
  Interventions: Other: follow up of cases fixed by posterior tension band plate

INTERVENTIONS:
Other: follow up of cases fixed by posterior tension band plate — Follow up of the reduction and functional outcome evaluation using the Majeed functional outcome score

SUMMARY:
The sacrum is the mechanical nucleus of the axial skeleton, serving as the base for the spinal column as well as the keystone for the pelvic ring.

Sacral fractures occur in approximately 45% of all pelvic fractures. the mechanism of injury resulting in sacral fractures typically is one of high energy from motor vehicle accidents and fall from a height.

Approximately 30% of sacral fractures are identified late. Unrecognized and inadequately treated sacral fractures may lead to painful deformity and progressive loss of neurological function. Delayed surgery for posttraumatic sacral deformity is complex, and the results are often less favorable than those of early surgery. Therefore, determination of an integrated diagnostic and therapeutic approach to sacral fractures should be a goal.

DETAILED DESCRIPTION:
Most sacral fractures can be treated non operatively. These include stable, non displaced sacral fractures without a significant associated pelvic ring disruption, fractures not involving the lumbosacral junction, and fractures without neurologic injury.

Surgical options range from minimally invasive techniques to formal open reduction and internal fixation. Techniques for neural decompression include laminotomy and foraminotomy, anterior bone disimpaction, and lumbosacral plexus neurolysis. Anterior sacral and pelvic stabilization techniques involve various methods of anterior stabilization of the pelvic ring (e.g., application of a sacroiliac plate). Posterior stabilization techniques include percutaneous sacroiliac screw fixation, bilateral sacroiliac screw fixation with posterior tension-band plate fixation, posterior alar plate fixation, and lumbopelvic segmental fixation.

Percutaneously placed iliosacral screws are commonly used for the fixation of sacroiliac joint disruptions and for sacral fractures. Adequate experience and intraoperative imaging is necessary to safely insert these screws, since the safe corridor for placement is fairly small. In some patients, such as those with a dysmorphic sacrum.

Transiliac posterior tension band fixation, offers an alternative method for stabilization of the posterior pelvic ring.

It is indicated in:vertically unstable comminuted sacral fractures, for which iliosacral screws may be insufficient. It is also indicated in patients with a dysmorphic sacrum in whom there is no safe corridor for placement of iliosacral screws. Threaded rods or a posterior plate may be secured to the posterior ilium.Also it can be used in bilateral sacral fracture; Late presented (neglected) sacral fractures and in osteoporotic sacral fracture.It is Minimally invasive technique with Less exposure to irradiation, image-independent, Easy, reproducible technique, Economic conventional implant and stable fixation.

ELIGIBILITY:
Inclusion Criteria:

* comminuted sacral fracture,
* bilateral sacral fracture,
* osteoporotic sacral fractures,
* spinopelvic dissociation and
* late presented (neglected) sacral fracture.

Exclusion Criteria:

* Patients with a preoperative diagnosis of a Morel- Lavallee lesion,
* unfit patients
* immature skeleton will be excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: fixation of sacral fractures by posterior tenstion band plate then follow up of the functional outcome by majeed outcome score at 6th month post operative
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Majeed functional outcome score | 6th month
  it is a pelvic injury-specific assessment divided into seven items such as pain, work, sitting, sexual intercourse, standing, gait unaided, and walking distance, with a total score range of 0-100 in order of decreasing disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut faculty of medicine, Asyut, Egypt

REFERENCES:
- [Background] Suzuki T, Hak DJ, Ziran BH, Adams SA, Stahel PF, Morgan SJ, Smith WR. Outcome and complications of posterior transiliac plating for vertically unstable sacral fractures. Injury. 2009 Apr;40(4):405-9. doi: 10.1016/j.injury.2008.06.039. Epub 2008 Dec 17. PMID 19095233
- [Background] Padalkar P, Pereira BP, Kathare A, Sun KK, Kagda F, Joseph T. Trans-iliosacral plating for vertically unstable fractures of sacral spine associated with spinopelvic dissociation: A cadaveric study. Indian J Orthop. 2012 May;46(3):274-8. doi: 10.4103/0019-5413.96376. PMID 22719112
- [Background] Sasso RC, Vaccaro AR, Chapman JR, Best NM, Zdeblick TA, Harris MB. Sacral fractures. Instr Course Lect. 2009;58:645-55. PMID 19385574